CLINICAL TRIAL: NCT01851161
Title: Pulmonary Tumor Motion Reduction and Improved Breathing Reproducibility by Prone Patient Positioning in Radiation Therapy
Brief Title: Prone Patient Positioning in Reducing Tumor Motion and Improving Breathing Reproduction in Patients With Lung Cancer Undergoing Radiation Therapy
Status: Terminated | Type: Observational
Why Stopped: Data analysis completed
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-12806; NCI-2013-00848 (Registry Identifier: NCI); HM12806 (Other: Virginia Commonwealth University IRB)
Record Dates: First submitted 2013-04-26; First posted 2013-05-10 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy; Radiation; Therapeutics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diagnostic (CT and 4D CT in supine and prone positioning): Patients undergo conventional CT scan and 4D CT scan in both supine and prone positioning before undergoing radiation therapy.
  Interventions: Procedure: computed tomography; Procedure: 4-dimensional computed tomography; Radiation: radiation therapy

INTERVENTIONS:
Procedure: computed tomography — Undergo conventional CT scan in both supine and prone positioning
  Other Names: tomography, computed
Procedure: 4-dimensional computed tomography — Undergo 4D CT scan in both supine and prone positioning
  Other Names: 4D-CT
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation, radiotherapy, therapy, radiation

SUMMARY:
This clinical trial studies prone patient positioning in reducing tumor motion and improving breathing reproduction in patients with lung cancer undergoing radiation therapy. Prone patient positioning during radiation therapy may help kill tumor cells without harming normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Quantify the three-dimensional tumor and normal tissue (thoracic and abdominal) motion, deformation and volume changes with the respiratory cycle during imaging in prone vs. supine positioning.

II. Quantify the three-dimensional tumor and normal tissue (thoracic and abdominal) motion, deformation and volume changes with the respiratory cycle and alterations thereof during a radiotherapy series.

OUTLINE:

Patients undergo one conventional computed tomography (CT) scan and one 4 dimensional CT (4D CT) scan in both supine and prone positioning before undergoing radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease on the planning computed tomography (CT) scan
* Patients with lung cancer visible on fluoroscopic imaging or planning CT who are scheduled to receive external beam radiation treatment will be eligible for this study

Exclusion Criteria:

* Patients requiring continuous supplemental oxygen due to the requirement of spirometry during all imaging studies
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General radiotherapy patient population during either the consultation or the simulation process. The possible participant will be contacted by either of the investigators or the study coordinator. Eligibility will be evaluated by observing the simulation data collected for each patient clinically, including any pretreatment fluoroscopy, digital simulation radiographs, cone beam CT, conventional or four-dimensional CT scans. Only clinical data will be used to assess eligibility. No extra imaging will be performed on a patient solely for the purpose of assessing eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2010-05; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Consistency of the respiratory pattern, quantified by the cycle-to-cycle variation in the respiration trace during imaging in prone vs. supine positioning | up to 90 days
  During the 4D CT patient respiration trace will be recorded using the RPM optical tracking device. The average and standard deviation of the amplitude, period, end of inhalation position, and end of exhalation position of the respiration trace will be calculated. Paired t tests and F tests will be used to evaluate differences between these quantities for supine and prone positioning.
Consistency of the respiratory pattern, quantified by the cycle-to-cycle variation in the respiration trace during a radiotherapy series | up to 90 days
  During the 4D CT patient respiration trace will be recorded using the RPM optical tracking device. The average and standard deviation of the amplitude, period, end of inhalation position, and end of exhalation position of the respiration trace will be calculated. Paired t tests and F tests will be used to evaluate differences between these quantities for supine and prone positioning.
Motion of the tumor and normal tissue evaluated in reference to the bony anatomy (vertebra) | up to 90 days
  The prone and supine image data acquired before the treatment onset will be used for planning. The computation of the doses will be performed on the dataset corresponding to the average position over the breathing pattern, based on previous studies indicating that a dose computation on this dataset approximates with sufficient accuracy the dose that will be received by the patient. The distributions of the tumor and normal tissue volumes in the prone and supine scans will be derived and the volume consistency will be assessed using the mean and the standard deviation of these distributions.

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Rosu, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Massey Cancer Center, Richmond, Virginia, United States